CLINICAL TRIAL: NCT06319274
Title: Efficacy and Safety of 72-hour Infusion of Prostacyclin (1 ng/kg/Min) in Mechanically Ventilated Patients With Infectious Pulmonary Endotheliopathy - a Multicenter Randomized, Placebo-controlled, Blinded, Investigator-initiated Trial
Brief Title: Infusion of Prostacyclin vs Placebo for 72-hours in Mechanically Ventilated Patients With Acute Respiratory Failure
Acronym: COMBAT-ARF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pär Johansson (Other)
Responsible Party: Sponsor-Investigator, Pär Johansson, Sponsor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMBAT-ARF
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Failure; Endothelial Dysfunction; Pulmonary Infection
Keywords: Endotheliopathy; SHINE
MeSH Terms: interventions — Iloprost; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomization active/placebo (1:1) parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) The preparation will be done by an unblinded study nurse independent of the including ICU´s, who will be responsible for preparing the investigational drug to be administered in a blinded fashion. Iloprost is a colorless fluid that is to be diluted in 0.9% saline. The infusion pump containing diluted active drug and placebo will be identical in both looks and behavior.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iloprost (Experimental): Patients randomized to active treatment (n=225 patients) will receive continuous infusion of iloprost for 72 hours after inclusion or until discharge to ward or death, whichever comes first.
  Interventions: Drug: Iloprost
- Isotonic saline (Placebo Comparator): Patients randomized to placebo treatment (n=225 patients) will receive continuous infusion of placebo for 72 hours after inclusion or until discharge to ward or death, whichever comes first.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Iloprost — Continuously infusion for 72 hours at 3 ml/hours. Treatment dose 1 ng/kg/min
  Other Names: Ilomedin
  Arms: Iloprost
Drug: Isotonic saline — Continuously infusion for 72 hours at 3 ml/hours
  Arms: Isotonic saline

SUMMARY:
The purpose of this clinical trial is to investigate the efficacy and safety of continuous intravenous administration of low dose iloprost versus placebo for 72-hours, in 450 mechanically ventilated patients with infectious respiratory failure. The study hypothesis is that iloprost may be beneficial as an endothelial rescue treatment as it is anticipated to deactivate the endothelium and restore vascular integrity in patients suffering from respiratory failure caused by endothelial breakdown, ultimately improving survival.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) is common in critically ill patients and 50% of all intensive care unit patients require mechanical ventilation. ARF occurs in a heterogenous patient group, most often in the setting of pneumonia, sepsis, aspiration of gastric contents or severe trauma and major surgery. Despite improvements in intensive care capabilities, ARF mortality remains high and the only treatment option, to date, is supportive care. A recent Cochrane analysis (2018) found no evidence for that any drug was effective in reducing deaths in mechanically ventilated patients with ARF, highlighting the high unmet medical need.

Given that the pulmonary system, apart from the brain, is the most highly vascularized vital organ in the body, extensive endothelial damage is a central feature of acute respiratory distress syndrome (ARDS) with respiratory failure being the rationale for the current study. Evidence support that iloprost infusion significantly improved endothelial function and integrity in mechanically ventilated patients with COVID-19 infection with reducing 28-day mortality by 50%.

The main objective in this clinical trial is to investigate whether continuous infusion of low dose iloprost at a dose of 1 ng/kg/min for 72-hours is safe and significantly reduce all-cause mortality at day 28.

Patients that are eligible for this trial will be temporarily incompetent due to acute severe illness relating to respiratory failure.

During the trial, patient will be given continuous infusion of low dose iloprost or placebo for 72 hours during their stay at the intensive care unit (ICU) and additional blood samples will be obtained at baseline, 24-, 48 and 72-hours.

This trial is conducted in accordance with the Helsinki 2 Declaration and International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use, Guideline for Good Clinical Practice (ICH-GCP) and in compliance with the protocol. As part of the quality assurance on-site monitoring visit will be performed by the an independent GCP-unit including source data verification. Standard Operation Procedure (SOP) will address protocol specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care patients (age ≥ 18 years)
* Suspected pulmonary infection
* Need for mechanical ventilation (< 24 hours from time of screening)
* soluble thrombomodulin (sTM) ≥ 4 ng/mL in blood plasma

Exclusion Criteria:

* Withdrawal from active therapy
* Pregnancy (non-pregnancy confirmed by patient having a negative urine- or plasma Choriogonadotropin (hCG) or being postmenopausal defined as females at 60 years old or beyond or at the investigators discretion)
* Septic shock according to the Sepsis 3 criteria AND a sTM> 10 ng/ml
* Known hypersensitivity to iloprost or to any of the other ingredients.
* Previously included in this trial or a prostacyclin trial within 30 days
* Life-threatening bleeding defined by the treating physician
* Known severe heart failure (NYHA class IV)
* Suspected acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | Day 28
  All-cause mortality at day 28

SECONDARY OUTCOMES:
90-day mortality | Day 90
  All-cause mortality at day 90
Vasopressor-free days | Until ICU discharge, maximun 90 days after randomization]
  Days alive without vasopressor in the ICU within 28- and 90 days
Renal replacement-free days | Until ICU discharge, maximun 90 days after randomization]
  Days alive without renal replacement in the ICU within 28- and 90 days
Mechanical ventilation free days | Until ICU discharge, maximun 90 days after randomization]
  Days alive without mechanical ventilation in the ICU within 28- and 90 days
Serious adverse reactions (SARs) | Until day 7 after randomization
  Total number and numbers of patient with one or more serious adverse reactions within the first 7 days
Serious adverse events (SAEs) | Until day 7 after randomization
  Total numbers and numbers of patients with one or more serious adverse events within the first 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Pär I Johansson, MD, DMSc, Study Director — Rigshospitalet, Denmark; Peter Soee-Jensen, MD, Principal Investigator — +4538682458
Locations (5):
- Denmark (5):
  - Dept. of Anaesthesia and Intensive Care, Bispebjerg Hospital, Copenhagen
  - Dept. of Intensive Care, Copenhagen University Hospital Herlev, Herlev
  - Dept. of Anaesthesia and Intensive Care, Nordsjaelands Hospital, Hillerød
  - Dept. of Intensive care, Hvidovre Hospital, Hvidovre
  - Department of Anesthesia and Intensive Care Medicine, Zealand University Hospital, Køge